CLINICAL TRIAL: NCT04109404
Title: Meningiomas and Treatment With CYPROTERONE ACETATE or Progestin: Retrospective Study in Patients Followed at the CHRU of Brest
Brief Title: Meningiomas and Treatment With CYPROTERONE ACETATE or Progestin
Acronym: MAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0030
Record Dates: First submitted 2019-09-23; First posted 2019-09-30 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Meningioma
Keywords: meningioma,; progestin,; cyproterone acetate
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators observe an increase risk of meningioma in patient treated by CYPROTERONE ACETATE or other form of progestin. Investigatorsdiscribe caractéristics of meningioma and treatement of the patients follow up in CHRU of Brest

DETAILED DESCRIPTION:
Retrospective study in CHRU of brest, the investigators selected patient with history of méningioma and treated by CYPROTERONE ACETATE, CHLORMADINONE ACETATE and NOMEGESTROL ACETATE essentially The investigators excluded patient with risk factor of meningioma added at hormonal treatment exposition The investigators discribe the caractéristique of patients: age, sex, duration of the treatment, the caractéristique of the meningioma: localization, grade, hormonal receptors, treatment by surgery or radiotherapy and changing after discontinuation of treatment

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years
* medical follow up in CHRU of Brest
* treated by CYPROTERONE ACETATE and/or CHLORMADINONE ACETATE NOMEGESTROL ACETATE, PROGESTERONE , DYDROGESTERONE PROMEGESTONE , NORETHISTERONE, LEVONORGESTREL , oestroprogestogenic contraception
* meningioma after treatement by progestin or CYPROTERONE ACETATE

Exclusion Criteria:

* history ofbreast cancer
* history of cerebral radiotherapy
* history of neurofibromatosis
* meningioma before treatement by progestin or CYPROTERONE ACETATE
* minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 6 men/110, 104 women/110 sex ratio 17.5:1 average duration of follow up: 5.5 years average age at diagnosis: 54 +/- 13 years
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of meningiomas caracteristics | 12 months
  meningiomas caracteristics in patient treated with CYPROTERONE ACETATE or Progestin description

SECONDARY OUTCOMES:
prescription status of progestogenic treatment | 12 months
  indications, duration of treatment, name and type of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Véronique KERLAN, PH, Principal Investigator — Service d'Endocrinologie-Diabétologie - CHRU de Brest
Locations (1):
- Département de Nutrition - CHRU de Brest, Brest, France

REFERENCES:
- [Background] Bernat AL, Oyama K, Hamdi S, Mandonnet E, Vexiau D, Pocard M, George B, Froelich S. Growth stabilization and regression of meningiomas after discontinuation of cyproterone acetate: a case series of 12 patients. Acta Neurochir (Wien). 2015 Oct;157(10):1741-6. doi: 10.1007/s00701-015-2532-3. Epub 2015 Aug 12. PMID 26264069
- [Background] S. Froelich, "Does cyproterone acetate promote multiple meningiomas?," 2009.